CLINICAL TRIAL: NCT05831436
Title: The Role of Licensing in Early Care and Education (TRLECE): Surveys Licensed Child Care Providers
Brief Title: The Role of Licensing in Early Care and Education: Licensed Providers
Acronym: TRLECE: LP
Status: Completed | Type: Observational
Sponsor: Child Trends (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); ICF International, Inc. (Unknown)
Responsible Party: Principal Investigator, Kelly Maxwell, Senior Scholar, Early Childhood Research, Child Trends
Other Study IDs: 17187003; 233201500034I-75P00119F37007 (Other Grant/Funding Number: OPRE, ACF, US Dept. Of Health and Human Services (HHSP))
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Child Care Providers Perceptions of the Licensing System
Keywords: Child care and early education; Child care licensing; Early care and education programs

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Child Trends, funded by the Office of Planning, Research, and Evaluation (OPRE), Administration for Children and Families (ACF) in the U.S. Department of Health and Human Services (HHS) will collect descriptive information for The Role of Licensing in Early Care and Education (TRLECE): Licensed Child Care Providers project. The goal of this information collection is to deepen the field's understanding of child care and early education licensing systems, which play a critical role in supporting positive outcomes for providers, families, and children. The investigators will conduct one round of survey data collection with a nationwide survey of licensed child care providers from all states.

DETAILED DESCRIPTION:
This study aims to advance understanding of the landscape of child care and early education licensing systems. State/territory child care and early education licensing agencies establish and monitor regulations that child care programs serving young children must meet to operate legally. These regulations and monitoring practices play a large role in the operations of child care programs but have received relatively little research attention. The field has limited information about features of state/territory licensing units and limited information about child care and early education providers' experiences and perceptions of licensing (i.e., there are a few findings from individual states but no national survey). Ultimately, TRLECE: Licensed Child Care Providers findings can inform changes to licensing policies and practices in the child care and early education field, guidance and technical assistance to state leaders, and future research.

The investigators will gather information for this descriptive study through a survey of licensed child care provider. This survey is designed to collect information about licensed child care and early education providers' experiences with child care licensing, including regulations and inspections; perceptions of the burden, value, and fairness of the licensing system; and perceived strengths of and challenges with the licensing system. The investigators intend to invite a stratified random sample of directors of center-based programs and family child care providers from all 50 states and the DC to participate and will aim to have 1,000 participants from each group.

ELIGIBILITY:
Inclusion Criteria:

* A randomly selected group of directors/owners/managers of licensed child care programs (providers) in all U.S. states and DC

Exclusion Criteria:

* Individuals who are not directors/owners/managers of licensed child care programs (providers) in all U.S. states and DC

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Licensed child care providers
Sampling Method: Probability Sample
Enrollment: 2884 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Child care provider survey | one time
  Survey developed by the study team to gather information regarding child care providers' overall perceptions of the licensing system (including value and burden), availability and utility of licensing information, perceptions of licensing staff and support, perceptions about components of the licensing system (including regulations, inspections, technical assistance, training, written guidance, licensing reports), strengths and challenges of the licensing system, areas for improvement, and demographic and program characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Kelly L Maxwell, PhD, Principal Investigator — Child Trends
Locations (1):
- Child Trends Headquarters, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared with the Child & Family Data Archive (CFData).
Time Frame: The team anticipates submitting IPD and supporting information to Child and Family Data Archive (CFData) roughly 6 months after the end of data collection. Data will be available after being reviewed by CFData. No end date on the availability of the data.
Access Criteria: Most data from the child care provider survey will be archived as public-use data with CFData and accessible on their website. Some data will be available as restricted-use only, following guidelines from CFData. Data will be shared with researchers for analyses related to the experiences and perceptions of licensed child care providers about the child care licensing system.